CLINICAL TRIAL: NCT00548561
Title: A Clinical Trial on TopotectTM (Dexrazoxane) in the Treatment of Accidental Extravasation of Anthracycline Anti-cancer Agents
Brief Title: Efficacy of TopotectTM (Dexrazoxane) for Accidental Extravasation of Anthracyclines
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TT01
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2013-11

CONDITIONS: Anthracycline Extravasation
Keywords: extravasation; anthracyclines
MeSH Terms: interventions — Dexrazoxane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dexrazoxane

SUMMARY:
The purpose of this study is to avoid surgical intervention following extravasation of anthracycline chemotherapy out of a vessel into the surrounding tissues.

DETAILED DESCRIPTION:
Accidental extravasation of anthracyclines including doxorubicin and its derivative epirubicin, may cause severe, progressive tissue necrosis requiring the surgical removal of any damaged tissue. Thus, the patient is subjected to major surgery causing substantial delay of the treatment of the primary cancer disease.

Tissue infiltration by anthracyclines may be detected by fluorescence microscopy. This test is performed at most hospitals in Denmark.

In a large preclinical trial, as well as 4 clinical cases, dexrazoxane has proven to prevent these severe tissue necroses. This trial will determine the effect of dexrazoxane as an acute treatment (acute antidote) in patients with anthracycline extravasation verified by fluorescence biopsy.

Purpose

Primary:

• To avoid surgical intervention following the accidental extravasation of anthracycline drug, and thus preventing the patient from sequelae.

Secondary:

* To avoid deleterious postponement of the cancer treatment itself.
* To evaluate and describe subjective and objective symptoms in the damaged area following treatment with TopotectTM.
* To evaluate tolerability/toxicity of TopotectTM used for this indication, according to the indicated schedule.

Trial Population 25 patients with accidental anthracycline extravasation confirmed by fluorescence microscopy

Trial Design Open-label clinical trial. Twenty-five consecutive patients with an acute (<6 hours) history of anthracycline extravasation confirmed by fluorescence microscopy (who in general practice are candidates for acute plastic surgical intervention) will be included.

Effect Variables Response rates, presence of late sequelae, time to progression, and clinical consequence of progression.

Safety Features

* Any toxicity caused by TopotectTM will be studied by blood tests, systematic questioning regarding subjective discomfort, as well as by objective clinical examination.
* A systematic clinical evaluation of the marked area of skin covering the area of extravasation will be performed to assure prompt treatment should any deterioration occur.
* Sequential colour photographs of the involved skin area will be taken.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients treated with anthracycline
2. Informed consent obtained from the patient.
3. Suspicion of anthracycline extravasation is defined as:

   A primary assessment by the physician on duty, which would activate the standard departmental procedure for treatment of anthracycline extravasation.

   The presence of at least one of the following:
   * pain
   * swelling
   * redness
4. The Topotect infusion must be started <6 hours after the accident.
5. The patient must be at least 18 years of age.
6. Performance status (PS) ≤2.
7. Suspicion of anthracycline extravasation from a central venous access device. -

Exclusion Criteria:

1. Known allergy towards dexrazoxane.
2. Reasonable suspicion of extravasation by other compounds than anthracyclines through the same intravenous access, e.g. vincristine, mitomycin, and vinorelbine, all of which may cause ulceration.
3. AST, ALT, bilirubin, LDH, serum alkaline phosphatase >3 x upper normal value
4. Neutropenia and thrombocytopenia ≥ CTC grade 2
5. Pregnant or nursing women
6. Women of childbearing age and potential, where the patient does not agree to use an efficient contraceptive (e.g. birth control pill or an intra-uterine device for 3 months previous to start of the trial medication or diaphragm plus a spermicide).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2001-06; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
The rate of surgical resection necessity by progressing necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Henning T Mouridsen, MD, Dr. med., Principal Investigator — Rigshospitalet, The Finsen Centre 5074, Blegdamsvej 9, DK-2100 Copenhagen
Locations (9):
- Denmark (9):
  - Aalborg Hospital South, Aalborg
  - Rigshospitalet, Copenhagen
  - Herlev County Hospital, Herlev
  - Herlev Hospital Hematological Department, Herlev
  - Herning District Hospital, Herning
  - Hilleroed Hospital, Hilleroed
  - Odense University Hospital, Odense
  - Roskilde County Hospital, Roskilde
  - Viborg Hospital, Viborg

REFERENCES:
- [Result] Mouridsen HT, Langer SW, Buter J, Eidtmann H, Rosti G, de Wit M, Knoblauch P, Rasmussen A, Dahlstrom K, Jensen PB, Giaccone G. Treatment of anthracycline extravasation with Savene (dexrazoxane): results from two prospective clinical multicentre studies. Ann Oncol. 2007 Mar;18(3):546-50. doi: 10.1093/annonc/mdl413. Epub 2006 Dec 21. PMID 17185744